CLINICAL TRIAL: NCT01406860
Title: Droperidol Versus Metoclopramide + Diphenhydramine for the Treatment of Primary Headaches in the Emergency Department: A Prospective Randomized, Double-blinded Trial.
Brief Title: Droperidol Versus Metoclopramide + Diphenhydramine for the Treatment of Primary Headaches
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment/drug shortages
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Brett A Faine, Clinical Pharmacy Specialist, University of Iowa
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201008798; University of Iowa
Record Dates: First submitted 2010-09-22; First posted 2011-08-01 (Estimated); Results first posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Primary Headaches (Includes Migraines, Tension, Cluster Headaches)
Keywords: Headaches; Migraines; Tension headaches; Cluster headaches
MeSH Terms: conditions — Cluster Headache; Headache; Migraine Disorders; Tension-Type Headache | interventions — Droperidol; Metoclopramide; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Droperidol (Experimental)
  Interventions: Drug: Droperidol
- Metoclopramide + Diphenhydramine (Active Comparator)
  Interventions: Drug: Metoclopramide + diphenhydramine

INTERVENTIONS:
Drug: Droperidol — Droperidol 1.25 mg IV x 1, may repeat 0.625 mg if needed at 60 minutes
  Arms: Droperidol
Drug: Metoclopramide + diphenhydramine — Metoclopramide 20 mg IV infusion q30 minutes as needed with a maximum of 4 doses + Diphenhydramine 25 mg IV injection x 1 given with the first dose of metoclopramide IV infusion and repeated x 1 given with the third metoclopramide IV infusion.
  Arms: Metoclopramide + Diphenhydramine

SUMMARY:
The purpose of this study is to determine if droperidol is equally as effective as metoclopramide for treatment of primary headaches in the Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old to 65 years old, diagnosis of primary headache

Exclusion Criteria:

* Allergy to study medications, pregnant, breast-feeding, prisoners, non-english speaking, not eligible to receive droperidol based on ED protocol (see below), patients in whom head trauma, infection, vascular disorders, and disorders of facial or cranial structures are suspected

ED Droperidol Protocol

Droperidol must NOT be used in patients with any of the following:

* Known or suspected QT prolongation, including congenital long QT syndrome
* Cardiac Disease [cardiomyopathy, congestive heart failure, hypertension, ischemic heart disease, myocardial infarction, bradycardia (< 50 bpm)]
* History of the following:

  * Renal failure
  * Cerebrovascular disease
  * Diabetes or hypoglycemia
  * Alcoholism/alcohol abuse
  * Pituitary insufficiency
  * Hypothyroidism
  * Hypothermia
  * Anorexia
* Advanced age (>65 yrs)
* Use of the following medications: digoxin, benzodiazepine, diuretics, IV opiates, or other medications known to prolong the QTc interval.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Van Heukelom, MD, Principal Investigator — University of Iowa; Christopher Hogrefe, MD, Principal Investigator — University of Iowa; Brett Faine, PharmD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Metoclopramide + Diphenhydramine: Metoclopramide: Metoclopramide 20 mg IV infusion q30 minutes as needed with a maximum of 4 doses + Diphenhydramine 25 mg IV injection x 1 given with the first dose of metoclopramide IV infusion and repeated x 1 given with the third metoclopramide IV infusion.
Period: Overall Study
Arm/Group | Droperidol | Metoclopramide + Diphenhydramine
Started | 11 | 8
Completed | 11 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Metoclopramide + Diphenhydramine: Metoclopramide: Metoclopramide 20 mg IV infusion q30 minutes as needed with a maximum of 4 doses.
  Diphenhydramine: Diphenhydramine 25 mg IV injection x 1 given with the first dose of metoclopramide IV infusion and repeated x 1 given with the third metoclopramide IV infusion.
- Total: Total of all reporting groups
Arm/Group | Droperidol | Metoclopramide + Diphenhydramine | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (9.01) | 30.6 (5.31) | 32.6 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Pain Scale (Numerical Rating Scale for Pain)
Description: Numerical Rating Scale for Pain on a scale of 0-10 with 10 representing the worst pain
Time Frame: Change in pain scores at 60 minutes from baseline as measured on the Numerical Rating Scale for Pain (NRS)
Population: Data were not collected
Arm/Group | Droperidol | Metoclopramide + Diphenhydramine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Length of Stay
Time Frame: Participants will be followed for the duration of their emergency department visit after the initiation of treatment (Average Length of stay in minutes)
Population: Data were not collected
Groups:
- Metoclopramide: Metoclopramide: Metoclopramide 20 mg IV infusion q30 minutes as needed with a maximum of 4 doses + Diphenhydramine 25 mg IV injection x 1 given with the first dose of metoclopramide IV infusion and repeated x 1 given with the third metoclopramide IV infusion.
Arm/Group | Droperidol | Metoclopramide
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: 24 Hour Pain Score
Description: 24 hour pain score (follow-up phone call)
Time Frame: 24 hours after discharge from ED
Population: Data were not collected
Arm/Group | Droperidol | Metoclopramide
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Adverse Effects
Description: Frequency of adverse effects in each arm
Time Frame: From the time when the treatment is initiated until the 24 hour follow-up phone survey
Population: Data were not collected
Arm/Group | Droperidol | Metoclopramide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Metoclopramide: Metoclopramide: Metoclopramide 20 mg IV infusion q30 minutes as needed with a maximum of 4 doses.
  Diphenhydramine: Diphenhydramine 25 mg IV injection x 1 given with the first dose of metoclopramide IV infusion and repeated x 1 given with the third metoclopramide IV infusion.
Arm/Group | Droperidol | Metoclopramide
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/8
Other Adverse Events (participants affected / at risk) | 0/11 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes